CLINICAL TRIAL: NCT02543554
Title: The Effect of Lung Protective Ventilation Initiated in the Emergency Department on the Incidence of Pulmonary Complications and Clinical Outcomes
Brief Title: ED Lung Protective Ventilation to Reduce Complications
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Brian Fuller, Associate Professor of Anesthesiology and Emergency Medicine, Washington University School of Medicine
Other Study IDs: 201409024
Record Dates: First submitted 2015-08-28; First posted 2015-09-07 (Estimated); Results first posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-05

CONDITIONS: Mechanical Ventilation; Ventilator-associated Conditions; ARDS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-intervention group: mechanically ventilated patients before implementation of ED lung protective ventilation
- Intervention group: mechanically ventilated patients after implementation of ED lung protective ventilation
  Interventions: Procedure: lung protective ventilation

INTERVENTIONS:
Procedure: lung protective ventilation — Lung protective ventilation strategy, which aims to deliver safe tidal volumes, appropriate PEEP, limit plateau pressure, and limit hyperoxia.
  Groups: Intervention group

SUMMARY:
Early mechanical ventilation, if delivered with injurious settings, can lead to pulmonary complications, such as acute respiratory distress syndrome (ARDS). Mechanical ventilation in the emergency department (ED) has been studied infrequently when compared to the intensive care unit; however, data suggests that ED-based mechanical ventilation has significant room for improvement and may also be a causative factor in ARDS incidence.

DETAILED DESCRIPTION:
This is a before-after study examining the impact of implementing lung protective ventilation in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated via an endotracheal tube in the ED

Exclusion Criteria:

* death in the ED,
* death or discontinuation of ventilation within 24 hours,
* chronic mechanical ventilation,
* ARDS while in the ED
* transfer to another hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients in the emergency department
Sampling Method: Probability Sample
Enrollment: 1705 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Fuller, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washinton University School of Medicine in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts BW, Mohr NM, Ablordeppey E, Drewry AM, Ferguson IT, Trzeciak S, Kollef MH, Fuller BM. Association Between Partial Pressure of Arterial Carbon Dioxide and Survival to Hospital Discharge Among Patients Diagnosed With Sepsis in the Emergency Department. Crit Care Med. 2018 Mar;46(3):e213-e220. doi: 10.1097/CCM.0000000000002918. PMID 29261567
- [Derived] Fuller BM, Ferguson I, Mohr NM, Stephens RJ, Briscoe CC, Kolomiets AA, Hotchkiss RS, Kollef MH. Lung-protective ventilation initiated in the emergency department (LOV-ED): a study protocol for a quasi-experimental, before-after trial aimed at reducing pulmonary complications. BMJ Open. 2016 Apr 11;6(4):e010991. doi: 10.1136/bmjopen-2015-010991. PMID 27067896

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pre-intervention Group | Intervention Group
Started | 1192 | 513
Completed | 1192 | 513
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-intervention Group | Intervention Group | Total
Number analyzed (Participants) | 1192 | 513 | 1705
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 754 | 357 | 1111
  >=65 years | 438 | 156 | 594
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (21.1) | 58.0 (24.0) | 58.8 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 564 | 210 | 774
  Male | 628 | 303 | 931
Region of Enrollment [Number; unit: participants]
  United States | 1192 | 513 | 1705

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Experience Pulmonary Complications After Admission From the Emergency Department
Time Frame: 7 days
Measure: Number; unit: participants
Groups:
- Pre-intervention Group: Before implementation of ED lung protection
- Intervention Group: after implementation of ED lung protective ventilation
Arm/Group | Pre-intervention Group | Intervention Group
Number analyzed (Participants) | 1192 | 513
participants | 171 | 38

2. Secondary Outcome: Number of Patients That Die During the Hospitalization
Time Frame: Patients will be followed for the duration of hospital stay
Measure: Number; unit: participants
Arm/Group | Pre-intervention Group | Intervention Group
Number analyzed (Participants) | 1192 | 513
participants | 338 | 105

ADVERSE EVENTS:
Arm/Group | Pre-intervention Group | Intervention Group
Serious Adverse Events (participants affected / at risk) | 0/1192 | 0/513
Other Adverse Events (participants affected / at risk) | 0/1192 | 0/513

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes